CLINICAL TRIAL: NCT04528719
Title: A Phase 1, Randomized, Observer-Blind, Placebo-Controlled, Dose Escalation Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1345, an mRNA Vaccine Targeting Respiratory Syncytial Virus (RSV), in Healthy Younger Adults Aged 18 to 49 Years, Women of Child-Bearing Potential Aged 18 to 40 Years, Healthy Older Adults Aged 65 to 79 Years, Japanese Older Adults Aged ≥ 60 Years, and RSV-Seropositive Children Aged 12 to 59 Months
Brief Title: A Dose Escalation Study to Evaluate Safety, Reactogenicity, and Immunogenicity of mRNA-1345 in Healthy Adults and in Children Who Are Respiratory Syncytial Virus (RSV)-Seropositive
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1345-P101
Record Dates: First submitted 2020-08-20; First posted 2020-08-27 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Respiratory Syncytial Virus
Keywords: Viral Diseases; Messenger RNA; Moderna; mRNA-1345; Respiratory syncytial virus; RSV Seropositive; Safety; Pediatric; Vaccines
MeSH Terms: conditions — Virus Diseases | interventions — mRNA-1345 respiratory syncytial virus vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For older adult Cohorts 7, 8, 9, 10, and 11, the second booster injection on Day 730 (Month 24) will be open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Cohort 1: Dose A in Younger Adults (Experimental): Single injection of Dose A of mRNA-1345 or matching-placebo on Day 1.
  Interventions: Biological: mRNA-1345; Drug: Placebo
- Cohort 2: Dose B in Younger Adults (Experimental): Single injection of Dose B of mRNA-1345 or matching-placebo on Day 1.
  Interventions: Biological: mRNA-1345; Drug: Placebo
- Cohort 3: Dose B in Younger Adults (Experimental): Three total injections, 1 injection of either Dose B of mRNA-1345 or matching-placebo per day on Day 1, Day 57, and Day 113.
  Interventions: Biological: mRNA-1345; Drug: Placebo
- Cohort 4: Dose C in Younger Adults (Experimental): Single injection of Dose C of mRNA-1345 or matching-placebo on Day 1.
  Interventions: Biological: mRNA-1345; Drug: Placebo
- Cohort 5: Dose D in Children (Experimental): Three total injections, 1 injection of either Dose D of mRNA-1345 or matching-placebo per day on Day 1, Day 57, and Day 113.
  Interventions: Biological: mRNA-1345; Drug: Placebo
- Cohort 6: Dose G in Children (Experimental): Three total injections, 1 injection of either Dose G of mRNA-1345 or matching-placebo per day on Day 1, Day 57, and Day 113.
  Interventions: Biological: mRNA-1345; Drug: Placebo
- Cohort 7: Dose A in Older Adults (Experimental): Two total injections, 1 injection of either Dose A of mRNA-1345 or matching-placebo per day on Day 1 and approximately 12 months later. Participants will receive second booster injection of Dose A of mRNA-1345 at Month 24.
  Interventions: Biological: mRNA-1345; Drug: Placebo
- Cohort 8: Dose B in Older Adults (Experimental): Two total injections, 1 injection of either Dose B of mRNA-1345 or matching-placebo per day on Day 1 and approximately 12 months later. Participants will receive second booster injection of Dose A of mRNA-1345 at Month 24.
  Interventions: Biological: mRNA-1345; Drug: Placebo
- Cohort 9: Dose C in Older Adults (Experimental): Two total injections, 1 injection of either Dose C of mRNA-1345 or matching-placebo per day on Day 1 and approximately 12 months later. Participants will receive second booster injection of Dose A of mRNA-1345 at Month 24.
  Interventions: Biological: mRNA-1345; Drug: Placebo
- Cohort 10: Dose E in Older Adults (Experimental): Two total injections, 1 injection of either Dose E of mRNA-1345 or matching-placebo per day on Day 1 and approximately 12 months later. Participants will receive second booster injection of Dose A of mRNA-1345 at Month 24.
  Interventions: Biological: mRNA-1345; Drug: Placebo
- Cohort 11: Dose F in Older Adults (Experimental): Two total injections, 1 injection of either Dose F of mRNA-1345 or matching-placebo per day on Day 1 and approximately 12 months later. Participants will receive second booster injection of Dose A of mRNA-1345 at Month 24.
  Interventions: Biological: mRNA-1345; Drug: Placebo
- Cohort 12: Dose E in Women of Child-Bearing Potential (Experimental): Single injection of Dose E of mRNA-1345 or matching-placebo on Day 1.
  Interventions: Biological: mRNA-1345; Drug: Placebo
- Cohort 13: Dose F in Women of Child-Bearing Potential (Experimental): Single injection of Dose F of mRNA-1345 or matching-placebo on Day 1.
  Interventions: Biological: mRNA-1345; Drug: Placebo
- Cohort 14: Dose A in Women of Child-Bearing Potential (Experimental): Single injection of Dose A of mRNA-1345 or matching-placebo on Day 1.
  Interventions: Biological: mRNA-1345; Drug: Placebo
- Cohort 15: Dose B in Japanese Older Adults (Experimental): Single injection of Dose B of mRNA-1345 or matching-placebo on Day 1.
  Interventions: Biological: mRNA-1345; Drug: Placebo

INTERVENTIONS:
Biological: mRNA-1345 — Formulation for injection
Drug: Placebo — 0.9% sodium chloride (normal saline) injection

SUMMARY:
The primary objectives of this study are to evaluate the tolerability and reactogenicity of a single injection of up to 5 dose levels of mRNA-1345 in younger adults, women of child-bearing potential, and older adults including Japanese older adults; of 3 injections of the middle dose level of mRNA-1345 given 56 days apart in younger adults; of a booster injection of mRNA-1345 given approximately 12 and 24 months after the primary injection in older adults; and of 3 injections of 1 of 2 dose levels of mRNA-1345 given 56 days apart in children who are RSV-seropositive.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy young adults ≥18 to ≤49 years of age, women of child-bearing potential ≥18 to ≤40 years of age, healthy older adults ≥65 to <80 years of age, Japanese older adults ≥ 60 years of age, and children ≥12 to < 60 months of age.
* Willing and physically able to comply with protocol-mandated follow-up, including all procedures.
* Adult participant or parent(s)/legal guardian(s) of pediatric participants has provided written informed consent for participation in this study, including all evaluations and procedures as specified by the protocol.

Specific inclusion criteria for adults (younger adults, women of child-bearing potential, and older adults [including Japanese older adults]):

* Has a body mass index (BMI) from ≥18 kilogram (kg)/meter (m)^2 to ≤35 kg/m^2.
* Female participants of non-child-bearing potential. This criterion does not apply for women of child-bearing potential Cohorts 12, 13, and 14.
* Female participants of child-bearing potential may be enrolled in the study, if the participant: 1) has a negative urine pregnancy test at Screening and on the day of vaccination; 2) has practiced adequate contraception or has abstained from all activities that could lead to pregnancy for 28 days prior to vaccination; 3) has agreed to continue adequate contraception through 3 months following the last injection; and 4) is not currently breastfeeding.

Specific inclusion criteria for children 12 to 59 months of age:

* Seropositive for RSV-neutralizing Abs at Screening.
* Has received routine immunizations appropriate for age per local guidance.
* Current height and weight above the third percentile for age.

Specific inclusion criteria for Japanese older adults:

* Japanese participants are defined as individuals born in Japan, with both parents and 4 grandparents who were born in Japan.

Key Exclusion Criteria:

* Has Screening laboratory values Grade ≥1 (younger adult, women of child-bearing potential, and pediatric participants) or >Grade 1 (older adult participants, including Japanese older adult participants).
* Is acutely ill or febrile on the day of the first injection.
* Has a significant medical history, including but not limited to:

  * Congenital or acquired immunodeficiency, including human immunodeficiency virus (HIV) infection.
  * Chronic hepatitis or suspected active hepatitis.
  * Bleeding disorder that is considered a contraindication to intramuscular (IM) injection or phlebotomy.
  * Dermatologic conditions that could affect local solicited AR assessments.
  * Any history of allergic or anaphylactic reactions following a vaccination that required medical intervention.
  * Autoimmune disease except for Hashimoto's disease.
  * Systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to the day of enrollment. Topical tacrolimus is allowed if not used within 14 days prior to the day of enrollment. Inhaled, nasal, and topical steroids are allowed.
  * Intravenous blood products (red cells, platelets, and immunoglobulins [Ig]) within 3 months prior to enrollment.
* Has received or plans to receive any licensed or authorized vaccine, to include COVID-19 vaccines, ≤ 28 days prior to the first injection (Day 1) or plans to receive a licensed vaccine within 28 days before or after any study vaccine injection, with the exception of licensed influenza vaccines, which may be received more than 14 days before or after any study vaccine injection. Nonstudy vaccinations should not be delayed.
* Has a history of myocarditis, pericarditis, or myopericarditis.

Specific exclusion criteria for older adults (Cohorts 7-11 and 15):

* Known history of poorly controlled hypertension (per determination of the Investigator) or systolic blood pressure >160 millimeters of mercury (mmHg) at the Screening visit.
* Known history of hypotension or systolic blood pressure <85 mmHg at the Screening visit.
* Poorly controlled diabetes mellitus (per determination of the Investigator).
* Diagnosis of significant chronic pulmonary disease (per determination of the Investigator) (such as, chronic obstructive pulmonary disease, asthma).
* Significant chronic cardiovascular disease (per determination of the Investigator).
* Resides in a nursing home.
* Anticipates the need for immunosuppressive treatment at any time during participation in the study.
* Diagnosis of malignancy within previous 10 years (excluding non-melanoma skin cancer and cervical carcinoma in-situ).

Specific exclusion criteria for children 12 to 59 months of age (Cohorts 5 and 6):

* Has received any monoclonal antibody at any time prior to Screening.
* Prior hospitalization for RSV disease in the last 2 years.
* Receipt of any prior systemic immunosuppressants or immune-modifying drugs.
* Any history of febrile seizures (inclusive of single simple febrile seizure).
* History of epilepsy.
* History of meningitis.

Ages: 12 Months to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 651 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Up to Day 737 (7 days after each injection)
Number of Participants with Unsolicited Adverse Events (AEs) | Up to Day 758 (28 days after the last injection)
Number of Participants with Serious AEs or Medically Attended AEs (MAAEs) | Up to Day 1095 (End of Study)

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) of Serum RSV Neutralizing and Binding Antibodies (Abs) | Up to Day 141 (Cohorts 5 and 6), up to Day 169 (Cohorts 1, 2, 4, 12, 13, 14, and 15), up to Day 281 (Cohort 3), and up to Day 1095 (Cohorts 7, 8, 9, 10, and 11)
Geometric Mean Fold-Rise of Postbaseline/Baseline Ab Titers | Up to Day 141 (Cohorts 5 and 6), up to Day 169 (Cohorts 1, 2, 4, 12, 13, 14, and 15), up to Day 281 (Cohort 3), and up to Day 1095 (Cohorts 7, 8, 9, 10, and 11)
Proportion of Participants with ≥2-fold and ≥4-fold Increases in Ab Titers from Baseline | Up to Day 141 (Cohorts 5 and 6), up to Day 169 (Cohorts 1, 2, 4, 12, 13, 14, and 15), up to Day 281 (Cohort 3), and up to Day 1095 (Cohorts 7, 8, 9, 10, and 11)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Paradigm Clinical Research Institute Inc - ClinEdge - PPDS, La Mesa, California
  - Mills Clinical Research, West Hollywood, California
  - Accel Research Site - Angel Kids Pediatrics - ERN - PPDS, DeLand, Florida
  - Accel Research Sites - Nona Pediatric Center - ERN - PPDS, Orlando, Florida
  - Palm Beach Research - ClinEdge - PPDS, West Palm Beach, Florida
  - Centricity Research - Roswell - HyperCore - PPDS, Columbus, Georgia
  - IResearch Atlanta LLC, Decatur, Georgia
  - Velocity Clinical Research (Savannah - Georgia) - PPDS, Savannah, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Synexus - Optimal Research - Peoria, Peoria, Illinois
  - Velocity Clinical Research (Sioux City - Iowa) - PPDS, Sioux City, Iowa
  - Michael W. Simon, M.D., PSC, Nicholasville, Kentucky
  - Velocity Clinical Research (Lafayette - Louisiana) - PPDS, Lafayette, Louisiana
  - Velocity Clinical Research (Metaire - Louisiana) - PPDS, Metairie, Louisiana
  - Velocity Clinical Research (Slidell - Louisiana) - PPDS, Slidell, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - Alliance for Multispecialty Research - Kansas City, Kansas City, Missouri
  - Velocity Clinical Research (Grand Island - Nebraska) - PPDS, Grand Island, Nebraska
  - Velocity Clinical Research (Hastings - Nebraska) - PPDS, Hastings, Nebraska
  - Velocity Clinical Research (Norfolk - Nebraska) - PPDS, Norfolk, Nebraska
  - Velocity Clinical Research (Omaha - Nebraska) - PPDS, Omaha, Nebraska
  - Velocity Clinical Research (Albuquerque - New Mexico) - PPDS, Albuquerque, New Mexico
  - Velocity Clinical Research (Binghamton - New York) - PPDS, Binghamton, New York
  - Velocity Clinical Research - Medford - ERN - PPDS, Medford, Oregon
  - Velocity Clinical Research - Columbia - PPDS, Columbia, South Carolina
  - Velocity Clinical Research (Greenville - South Carolina) - PPDS, Greenville, South Carolina
  - Cyfair Clinical Research Center - ERN - PPDS, Houston, Texas
  - Flourish Research - San Antonio - PPDS, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Tanner Clinic, Layton, Utah
  - Clinical Research Partners LLC, Richmond, Virginia

REFERENCES:
- [Derived] Schnyder Ghamloush S, Fanning S, Essink B, Eder F, Snape MD, Stoszek SK, Guo R, Dhar R, Righi V, Morsy L, Kapoor A, El Asmar L, Shaw CA. Safety and immunogenicity of an mRNA-based RSV vaccine in seropositive children aged 12-59 months. Hum Vaccin Immunother. 2025 Dec;21(1):2557676. doi: 10.1080/21645515.2025.2557676. Epub 2025 Sep 15. PMID 40953212
- [Derived] Fitz-Patrick D, Mihara H, Mills A, Mithani R, Kapoor A, Dhar R, Wilson L, Guo R, Simorellis AK, Panozzo CA, Reuter C, Wilson E, Chen GL, Stoszek SK, Shaw CA, Goswami J. Safety and immunogenicity of an mRNA-based RSV vaccine in Japanese older adults aged >/=60 years: A phase 1, randomized, observer-blind, placebo-controlled trial. Respir Investig. 2024 Nov;62(6):1037-1043. doi: 10.1016/j.resinv.2024.08.011. Epub 2024 Sep 9. PMID 39255587
- [Derived] Shaw CA, Essink B, Harper C, Mithani R, Kapoor A, Dhar R, Wilson L, Guo R, Panozzo CA, Wilson E, Simorellis AK, Reuter C, Stoszek SK, Chen GL, Das R, Goswami J. Safety and Immunogenicity of an mRNA-Based RSV Vaccine Including a 12-Month Booster in a Phase 1 Clinical Trial in Healthy Older Adults. J Infect Dis. 2024 Sep 23;230(3):e647-e656. doi: 10.1093/infdis/jiae081. PMID 38385566
- [Derived] Shaw CA, Mithani R, Kapoor A, Dhar R, Wilson L, El Asmar L, Schnyder-Ghamloush S, Schaefers K, August A, Stoszek SK, Chen GL. Safety, Tolerability, and Immunogenicity of an mRNA-Based Respiratory Syncytial Virus Vaccine in Healthy Young Adults in a Phase 1 Clinical Trial. J Infect Dis. 2024 Sep 23;230(3):e637-e646. doi: 10.1093/infdis/jiae035. PMID 38298125